CLINICAL TRIAL: NCT02773056
Title: Prosthetic Socket Interface Design on Socket Comfort, Residual Limb Health, and Function for the Transfemoral Amputee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00021886; CDMRP-MR140125 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2015-12-08; First posted 2016-05-16 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Amputation
Keywords: transfemoral; amputation; perspiration; socket; socket comfort

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Socket 1 (Ischial Ramus Containment) (Active Comparator): This arm included unilateral transfemoral amputees who were assessed while using the Ischial Ramus Containment socket.
  Interventions: Device: Ischial Ramus Containment (IRC)
- Socket 2 (Dynamic Socket IRC) (Active Comparator): This arm included unilateral transfemoral amputees who were assessed while using the Dynamic Socket Ischial Ramus Containment socket.
  Interventions: Device: Dynamic Socket Ischial Ramus Containment (IRC)
- Socket 3 (Sub-Ischial Interface) (Active Comparator): This arm included unilateral transfemoral amputees who were assessed while using the Sub-Ischial Interface socket.
  Interventions: Device: Sub-Ischial Interface (Sub-I)

INTERVENTIONS:
Device: Ischial Ramus Containment (IRC) — Ischial Ramus Containment (IRC) is the standard of care socket
  Arms: Socket 1 (Ischial Ramus Containment)
Device: Dynamic Socket Ischial Ramus Containment (IRC) — Dynamic Socket Ischial Ramus Containment (IRC) is a comparator study socket
  Arms: Socket 2 (Dynamic Socket IRC)
Device: Sub-Ischial Interface (Sub-I) — Sub-Ischial Interface (Sub-I) is a comparator study socket
  Arms: Socket 3 (Sub-Ischial Interface)

SUMMARY:
The primary objective of this clinical trial is to determine if the Dynamic Socket and Sub-Ischial alternative interface designs improve socket comfort, residual limb health, increase function and be preferred over the standard of care Ischial Ramus Containment (IRC) interface for the military and veteran living with transfemoral limb loss.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral above the knee amputees of non-dysvascular etiology
* 100-275 lbs
* ≥ 1 yr. of prosthetic experience
* Independent community ambulator
* Self-reported ability to walk for 20min consecutively

Exclusion Criteria:

* Above the knee amputees of dysvascular etiologies
* Body weight <100 or >275 lbs
* Does not speak English or Spanish
* Use of an assistive device (i.e. canes, walkers)
* Transtibial, hip disarticulation, hemipelvectomy, partial foot and bilateral amputees
* Known skin issues
* Known cognitive impairment

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Skin Temperature | Accommodation with new prosthetic sockets is approximately 10 days
  Continuous skin temperature measurement (Celsius) will be taken during treadmill walking at self-selected comfortable speed
Perspiration | Accommodation with new prosthetic sockets is approximately 10 days
  Perspiration will be measured by tare weight (grams) following treadmill walking.
Vertical Interface Movement (Pistoning) | Accommodation with new prosthetic sockets is approximately 10 days
  Pistoning will be defined as the numerical difference of interface to skeletal movement (cm) between simulated swing (lifting the prosthetic side) and stance (single support on the prosthetic side) as measured by coronal X-Ray.

SECONDARY OUTCOMES:
Balance and Stability | Accommodation with new prosthetic sockets is approximately 10 days
  The gold standard test of standing balance is the sensory organization test (SOT) administered on the Neurocom Equitest platform. The SOT score is a unitless number. Subjects stand on a pair of platforms that record force data and tilt in the sagittal plane during 6 varying conditions that challenge the visual, vestibular and somatosensory systems. With compromised ability to use an ankle strategy for balance, a hip strategy is routinely adopted, therefore higher interface trim lines could adversely affect performance on this test.
Comfort | Accommodation with new prosthetic sockets is approximately 10 days
  The Socket Comfort Score (rated on an 11-point 0-10 scale) will be used to assess patients' comfort in the respective sockets.
Preference | Accommodation with new prosthetic sockets is approximately 10 days
  Patients will be asked which socket they preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Highsmith, PhD, CP, PT, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kahle JT, Miro RM, Ho LT, Porter MR, Lura DJ, Carey SL, Lunseth P, Swanson AE, Highsmith MJ. Effect of transfemoral prosthetic socket interface design on gait, balance, mobility, and preference: A randomized clinical trial. Prosthet Orthot Int. 2021 Aug 1;45(4):304-312. doi: 10.1097/PXR.0000000000000013. PMID 33856157